CLINICAL TRIAL: NCT01937065
Title: Social Deprivation and Initial Presentation of 12 Cardiovascular Diseases: a CALIBER Study
Acronym: IP4
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Harry Hemingway, Professor, University College, London
Other Study IDs: 12_153R_IP4
Record Dates: First submitted 2013-07-02; First posted 2013-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Abdominal Aortic Aneurysm; Coronary Heart Disease NOS; Unheralded Corronary Death; Intracerebral Haemorrhage; Heart Failure; Ischemic Stroke; Myocardial Infarction; Stroke; Peripheral Arterial Disease; Stable Angina Pectoris; Subarachnoid Haemorrhage; Transient Ischemic Attack; Unstable Angina; Cardiac Arrest, Sudden Cardiac Death
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Cerebral Hemorrhage; Heart Failure; Ischemic Stroke; Myocardial Infarction; Stroke; Peripheral Arterial Disease; Angina, Stable; Subarachnoid Hemorrhage; Ischemic Attack, Transient; Angina, Unstable; Heart Arrest; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment
  Interventions: Other: No treatment

INTERVENTIONS:
Other: No treatment

SUMMARY:
Study of heterogeneity in associations between social deprivation and the initial presentation of 12 cardiovascular diseases.

DETAILED DESCRIPTION:
This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

ELIGIBILITY:
Inclusion Criteria:

* One year prior to study entry (up-to-standard follow-up, CPRD quality research standard).
* 30 years or older
* Recorded sex
* Free of symptomatic CVD at inclusion.

Exclusion Criteria:

* Pregnant women in the 6 months before the eligibility date

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1,93 million patients registered in Clinical Practice Research Datalink (CPRD) practices
Sampling Method: Non-Probability Sample
Enrollment: 1937360 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Hazard ratios for the associations between social deprivation and initial presentation of 12 cardiovascular diseases. | Followed for the duration of general practice registration between January 1997 and March 2010, an expected average of 5 years
  Associations studied:
  * overall
  * by sex
  * by age group
  * in high risk groups (smokers, hypertensive disease, obese, diabetic, depression)
  * before and after the introduction of the Quality and Outcomes Framework in England

SECONDARY OUTCOMES:
Lifetime cumulative incidence per quintile of social deprivation | Followed for the duration of general practice registration between January 1997 and March 2010, an expected average of 5 years

OTHER OUTCOMES:
Heterogeneity in associations across 12 cardiovascular diseases using the Tau-squared statistic and I-square statistics. | Followed for the duration of general practice registration between January 1997 and March 2010, an expected average of 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

REFERENCES:
- See also: Related Info — https://www.caliberresearch.org/